CLINICAL TRIAL: NCT01714674
Title: The Impact of Dietary Nitrate Supplementation on Exercise-induced Cardiac Troponin T Release in Type 2 Diabetic Patients
Brief Title: Nitrate and Exercise-induced Cardiac Troponin T in Type 2 Diabetes
Acronym: NO troponin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: METC 12-3-033; NL41071.068.12 (Other: ccmo)
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2012-11-01 (Estimated); Status verified 2012-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: cardiac troponin T; cTnT; exercise; dietary nitrate
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiomyopathy, Familial Restrictive, 3; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo beverage (Placebo Comparator): the impact of placebo (no active substance) on exercise-induced cTnT release
  Interventions: Dietary Supplement: NaCl beverage
- Dietary nitrate beverage (Active Comparator): The impact of dietary nitrate (active substance) on exercise-induced cTnT release
  Interventions: Dietary Supplement: Dietary nitrate beverage

INTERVENTIONS:
Dietary Supplement: Dietary nitrate beverage — ingestion of single dose NaNO3 beverage two hours prior to exercise bout
  Arms: Dietary nitrate beverage
Dietary Supplement: NaCl beverage — ingestion of single dose NaCl beverage two hours prior to exercise bout
  Arms: Placebo beverage

SUMMARY:
Blood cardiac troponin T (cTnT) concentration is a widely used marker of acute cardiac injury. Previous research has shown that type 2 diabetic patients may experience large increments in cTnT levels over the subsequent hours following a single bout of moderate-intensity endurance-type exercise. This phenomenon is likely attributed to cardiac ischemia-reperfusion injury caused by reduced nitric oxide (NO) bioavailability. Recent evidence indicates that ingestion of dietary nitrates dramatically increases the bioavailability of NO, and as such, may be protective against cardiac ischemia-reperfusion injury.

The investigators hypothesize that dietary nitrate supplementation blunts the rise in cTnT levels following exercise in type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* exercise-induced cTnT release (>3ng/L)

Exclusion Criteria:

* HbA1c <6.0% or >10.0%
* morbid obesity (BMI>35 kg/m2)
* incident cardiovascular events in the last year (heart attack, stroke
* use medication which contain nitrates and/or having vasodilatory effects

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2012-10; Primary Completion 2013-03 (Estimated); Study Completion 2013-05 (Estimated)

PRIMARY OUTCOMES:
Cardiac troponin T | 9 hours, hourly time intervals
  Cardiac troponin T levels will be assessed before exercise and over the 6-hour period following a single session of exercise.

SECONDARY OUTCOMES:
Plasma nitrate | 9 hours, hourly time intervals
  Cardiac troponin T levels will be assessed before exercise and over the 6-hour period following a single session of exercise.
Plasma nitrite | 9 hours, hourly time intervals
  Plasma nitrite levels will be assessed before exercise and over the 6-hour period following a single session of exercise.
Blood pressure | day
  Blood pressure will be measured various time during the day.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, PhD, Principal Investigator — Maastricht UMC
Locations (1):
- Maastricht UMC, Maastricht, Netherlands

REFERENCES:
- See also: research unit — http://www.m3-research.nl/